CLINICAL TRIAL: NCT05524103
Title: A Phase Ⅰ, Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of ALMB-0166 in Patients With Acute Spinal Cord Injury
Brief Title: Study to Evaluate the Safety and Pharmacokinetics of ALMB-0166 in Patients With Acute Spinal Cord Injury
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AlaMab Therapeutics (Shanghai) Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALMB-0166-CN-101
Record Dates: First submitted 2022-08-26; First posted 2022-09-01 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2022-08

CONDITIONS: Acute Spinal Cord Injury

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ALMB-0166 (Experimental): Two-thirds of patients will be randomized to receive a single dose of ALMB-0166 within 72 hours after spinal cord injury.
  Interventions: Drug: ALMB-0166
- Placebo (Placebo Comparator): One-third of patients will be randomized to receive a single dose of placebo within 72 hours after spinal cord injury.
  Interventions: Drug: ALMB-0166

INTERVENTIONS:
Drug: ALMB-0166 — A single dose of ALMB-0166 injection.
  Other Names: ALMB 0166

SUMMARY:
The purpose of this study is to assess the safety, tolerability and pharmacokinetics of ALMB-0166 in patients with acute spinal cord injury.

DETAILED DESCRIPTION:
This is a phase 1, randomized, double-blinded, placebo-controlled, single ascending dose study to evaluate the safety, tolerability and pharmacokinetics of ALMB-0166 in patients with acute spinal cord injury.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18-75 years old.
* ASIA (American Spinal Injury Association) impairment scale grade B or C.
* Spinal cord injury at the cervical and thoracic level (C4-T12).
* Scheduled to undergo a spinal surgery within 72 hours after the initial injury.
* Acute spinal cord injury that requires surgery as judged by the investigator.
* Ability to understand the entire process of this study, voluntarily participate and sign written informed consent form.
* Female patients with childbearing potential must have a negative serum pregnancy test and must be non-lactating. Male patients with female partners of childbearing age and female patients in childbearing age must use a medically approved contraceptive method during the study period and for 3 months after the administration. Male patients must avoid donating sperm during the study period.

Exclusion Criteria:

* Surgical treatment is not necessary or impossible according to the judgment of the investigator or for other reasons.
* Penetrating spinal cord injury or complete spinal cord rupture.
* Accompanying traumatic brain injury (TBI) with visible structural lesions or diagnostic images, such as intracranial hemorrhage.
* Patients with acute and chronic diseases that have caused neurological deficits (e.g., multiple sclerosis, Guillain-Barré syndrome, etc.)
* Body temperature is lower than 35℃.
* Patients with hemoglobin level <90 g/L.
* Difficulty in completing the study due to coma, mental illness or other reasons.
* History of drug abuse or dependence.
* Allergies to macromolecular drugs or a previous history of severe drug allergies.
* Positive serology for HIV and syphilis or active Hepatitis B or Hepatitis C.
* History of serious diseases of other organ systems such as heart, lungs, liver, or kidneys, who are judged by the investigator to be unsuitable to participate in clinical trials; for example, cardiovascular disease such as New York Heart Association (NYHA) Grade II or higher congestive heart failure, unstable angina pectoris, myocardial infarction, etc., and pulmonary fibrosis or interstitial lung disease, etc. within 6 months before the administration.
* Patients with active malignant tumour, or a history of treatment for invasive tumours within 3 years. Patients with stage I tumours who have received definite local treatments and are considered unlikely to recur can be accepted. Patients with a history of treatment for carcinoma in situ (such as non-invasive) and a history of non-melanoma skin cancer can be accepted.
* Participated in other clinical trials and received drug treatment within 30 days before enrolment.
* Patients with contraindications to lumbar puncture.
* Any other issue which, in the opinion of the investigator, made the patient unsuitable for study participation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-04-15 (Actual); Primary Completion 2025-02-08 (Actual); Study Completion 2025-02-08 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events of ALMB0166 [Safety and Tolerability] | Up to 2 months post-dose
  Assessment of the safety and tolerability of single dose of ALMB-0166

SECONDARY OUTCOMES:
Maximum Plasma Concentration [Cmax] of ALMB0166 | Pre-dose and multiple timepoints up to 2 months post-dose
  Assessment of pharmacokinetic (PK) profile
Assessment of anti-drug antibodies (ADA) | Pre-dose and multiple timepoints up to 2 months post-dose
  Assessment of anti-drug antibodies (ADA)
Assessment of American Spinal Cord Injury Association (ASIA) sensory, motor and injury grading. | Up to 2 months post-dose
  Sensory score range: 0-224 points; Sports score range: 0-100 points; Classification range: A-E. Higher scores mean a better outcome.
Assessment of Short-form Visual Analogue Scale (VAS) | Up to 2 months post-dose
  Scoring range: 0-10 points. Higher scores mean a worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Tian Jiali, Doctor, Principal Investigator — Peking Union Medical College
Locations (2):
- China (2):
  - Peking University Third Hospital Medical Science Research Ethic Committee, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: No